CLINICAL TRIAL: NCT02304016
Title: Evaluation of the Effect of Pelvic Floor Physical Therapy on Patients With 3rd and 4th Degree Obstetrical Lacerations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Boston Urogynecology Associates (Other)
Responsible Party: Principal Investigator, Eman Elkadry, M.D., Clinical Instructor, Boston Urogynecology Associates
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014P000141
Record Dates: First submitted 2014-11-26; First posted 2014-12-01 (Estimated); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Obstetrical Lacerations; Obstetric; Injury Pelvic Floor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pelvic floor physical therapy (Experimental)
  Interventions: Behavioral: Pelvic floor physical therapy
- Observatoin (No Intervention)

INTERVENTIONS:
Behavioral: Pelvic floor physical therapy — Patients in this arm will be receiving pelvic floor physical therapy
  Arms: Pelvic floor physical therapy

SUMMARY:
The purpose of this study is to determine if patients with third and fourth degree obstetric lacerations benefit from a short course of pelvic floor physical therapy in the immediate postpartum period.

DETAILED DESCRIPTION:
The proposed study is a prospective, randomized pilot trial. We aim to answer the question: do patients with third and fourth degree obstetric lacerations benefit from a short course pelvic floor physical therapy in the immediate postpartum period?

Forty patients experiencing third or fourth degree obstetric laceration at either BIDMC or Mount Auburn Hospital will be identified and randomized in a 1:1 ratio. Half of the patients will receive a 10-12 week course of pelvic floor physical therapy at Marathon PT to begin one to two weeks postpartum. Those assigned to the control will not receive pelvic floor physical therapy which is the current standard of care. They will also agree not to seek pelvic floor physical therapy during until at least 14 weeks postpartum without discussing with study investigators. At 14 weeks postpartum they will be offered pelvic floor physical therapy. At 1-2 weeks postpartum, 6-8 weeks postpartum, and 12-14 weeks postpartum, all study subjects will complete the Pelvic Floor Impact Questionnaire - 7 (PFIQ-7), the Pelvic Floor Distress Inventory - 20 (PFDI-20), the Female Sexual Function Index (FSFI), the Patient Global Impression of Severity (PGI-S) Scale and the Patient Global Impression of Improvement (PGI-I) Scale all of which are validated surveys. Surveys will be completed online via REDCap using computers at Marathon PT for treatment group subjects and at home or in a location of their choosing for control subjects. Control patients will be given the option of beginning pelvic floor PT after 14 weeks postpartum. Should they decide to pursue pelvic floor PT at that time, they will have the option to continue to fill out periodic surveys via REDCap, but will not be required to do so.

ELIGIBILITY:
Inclusion Criteria:

* Vaginal delivery at either BIDMC or Mt. Auburn Hospital complicated by either third or fourth degree perineal laceration
* Age 18 or older

Exclusion Criteria:

* History of previous vaginal delivery after 24 weeks gestation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-12; Primary Completion 2020-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Improvement in pelvic floor function (change in PFDI-20) | 12-24 weeks
  The primary outcome will be the change in PFDI-20 from baseline to the final assessment at approximately 12-24 weeks postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Eman Elkadry, MD, Principal Investigator — Harvard Medical School (HMS and HSDM)
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Mount Auburn Hospital, Cambridge, Massachusetts

REFERENCES:
- [Derived] Von Bargen E, Haviland MJ, Chang OH, McKinney J, Hacker MR, Elkadry E. Evaluation of Postpartum Pelvic Floor Physical Therapy on Obstetrical Anal Sphincter Injury: A Randomized Controlled Trial. Female Pelvic Med Reconstr Surg. 2021 May 1;27(5):315-321. doi: 10.1097/SPV.0000000000000849. PMID 32282525